CLINICAL TRIAL: NCT03151434
Title: Randomized Prospective Study Comparing Paravertebral Catheters, Single Shot Paravertebral Block, Thoracic Epidural, for Postoperative Analgesia Following Video-assisted Thoracoscopic Surgery
Brief Title: Comparison of Three Different Pain Blocks for Subjects Undergoing VATS (Video Assisted Thoracoscopic Surgery) Procedure.
Acronym: VATS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yar Yeap, Director, Acute Pain Service Assistant Professor of Clinical Anesthesiology Indiana University School of Medicine Department of Anesthesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1601583558
Record Dates: First submitted 2017-03-22; First posted 2017-05-12 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Video Assisted Thoracoscopic Surgery; Pain, Postoperative; Pain, Acute
Keywords: VATS; pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Pain | interventions — Tea; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Patients randomized to epidural, single shot paravertebral block, and paravertebral catheter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group #1 (Active Comparator): US Guided Single Shot Paravertebral Block
  Interventions: Drug: US Guided Single Shot Paravertebral Block (0.2% ropivicaine infusion)
- Group #2 (Active Comparator): US Guided Paravertebral Catheter
  Interventions: Drug: US Guided Paravertebral Catheter (0.2% ropivicaine bolus)
- Group #3 (Active Comparator): Thoracic Epidural
  Interventions: Drug: Thoracic Epidural (0.125% bupivicaine/hydromorphone)

INTERVENTIONS:
Drug: US Guided Single Shot Paravertebral Block (0.2% ropivicaine infusion) — Single shot paravertebral block will be placed under ultrasound guidance at the thoracic region prior to surgery.
  Other Names: US Guided Single Shot Paravertebral Block
  Arms: Group #1
Drug: US Guided Paravertebral Catheter (0.2% ropivicaine bolus) — Paravertebral catheter will be placed under ultrasound guidance at the thoracic region prior to surgery.
  Other Names: US Guided Paravertebral Catheter
  Arms: Group #2
Drug: Thoracic Epidural (0.125% bupivicaine/hydromorphone) — Epidural catheter will be placed in the thoracic region prior to surgery.
  Arms: Group #3

SUMMARY:
The purpose of this study is to compare three different pain control methods on subjects who are scheduled to undergo VATS (video-assisted thoracoscopic surgery) procedures. The study will compare their pain scores, narcotic needs, patient satisfaction scores, and narcotic side effects.

DETAILED DESCRIPTION:
All patients will be consented on the morning of surgery. All the thoracic epidurals and ultrasound-guided paravertebral blocks will be placed preoperatively. The procedures will be done using sterile technique with masks, hats, and sterile gloves. All procedures will be placed under the supervision of the attending anesthesiologist on the acute pain service or the attending anesthesiologist in the operating room.

Thoracic epidurals will be placed using the Arrow thoracic epidural kit. The epidural will be placed at the appropriate level to cover the entry site for the VATS procedure. Placement will be determined by anatomical landmarks. The epidural needle will be advanced toward the epidural space utilizing a Paramedian approach and loss-of-resistance technique. A sterile catheter will then be secured in place and the epidural infusion will be started at the end of the case.

Ultrasound guided paravertebral catheter and single shot paravertebral block will be accomplished using an ultrasound transducer at the thoracic level. This will be done using an in-plane or out-of-plane approach, at the discretion of the anesthesia staff performing the procedure. Then a needle will be inserted the needle into the paravertebral space and local anesthetic injected. Then a catheter will be placed within the injectate and secured in place in the case of the paravertebral catheter. The 0.2% Ropivicaine will be delivered by OnQ pump.

General anesthesia will be induced and the patient will be placed in the lateral position for the VATS procedure. The patients will be intubated with dual lumen endotracheal tubes and placed on one-lung ventilation for the procedure.

All patients will receive intravenous patient-controlled analgesia (PCA hydromorphone) post-operatively for breakthrough pain. They will also be scheduled on PO acetaminophen. PO oxycodone PRN will be started on POD 1 once patients tolerate diet.

Opioid usage at 1,24,48,72 hours after the block will be recorded by a member of the research team. Pain scores at rest and on movement (knee flexion) will be measured by the investigator using Visual Analog Scale (VAS). Nausea will be measured using a categorical scoring system (none=0; mild=1; moderate=2; severe=3). Sedation scores will also be assessed by a member of the study team using a sedation scale (awake and alert=0; quietly awake=1; asleep but easily roused=2; deep sleep=3). All these parameters will be measured at 1, 24, 48 and 72 hours after the epidural or PVB. Patients will be encouraged to ambulate on postoperative day 1 under supervision.

All catheters will be removed by APS (Acute Pain Service) while patients are still in the hospital. APS will continue to follow the patients until catheter removal. Patient's hospital length of stay and readmission rate will be recorded from NSQIP (National Surgical Quality Improvement Program) data.

All patients will receive a phone call 6 months after surgery for assessment for chronic post-surgical pain. Patients will be assessed by a member of the research team over the phone. They will be assessed on their pain score and narcotic usage by using the Brief Pain Inventory. Study participation will conclude after the 6 month follow questionnaire has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Pt undergoing VATS procedure at Indiana University Hospital
* ASA 1,2,3 or 4
* Age 18 or older, male or female
* Desires Regional anesthesia for postoperative pain control

Exclusion Criteria:

* Any contraindication for Thoracic Epidural or Paravertebral block
* History of substance abuse in the past 6 months
* Patient staying intubated after surgery
* Known allergy or other contraindications to the study medications , which include dilaudid, bupivacaine, ropivacaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University Hospital
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bottiger BA, Esper SA, Stafford-Smith M. Pain management strategies for thoracotomy and thoracic pain syndromes. Semin Cardiothorac Vasc Anesth. 2014 Mar;18(1):45-56. doi: 10.1177/1089253213514484. Epub 2013 Dec 12. PMID 24336691
- [Background] Daly DJ, Myles PS. Update on the role of paravertebral blocks for thoracic surgery: are they worth it? Curr Opin Anaesthesiol. 2009 Feb;22(1):38-43. doi: 10.1097/ACO.0b013e32831a4074. PMID 19237975
- [Background] Dango S, Harris S, Offner K, Hennings E, Priebe HJ, Buerkle H, Passlick B, Loop T. Combined paravertebral and intrathecal vs thoracic epidural analgesia for post-thoracotomy pain relief. Br J Anaesth. 2013 Mar;110(3):443-9. doi: 10.1093/bja/aes394. Epub 2012 Nov 14. PMID 23151421
- [Background] Davies RG, Myles PS, Graham JM. A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy--a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2006 Apr;96(4):418-26. doi: 10.1093/bja/ael020. Epub 2006 Feb 13. PMID 16476698
- [Background] El-Morsy, W. Z. (2013). Thoracic epidural analgesia versus parenteral morphine for post-thoracotomy pain relief. Ain-Shams Journal of Anaesthesiology, 6(2), 180.
- [Background] Fortier S, Hanna HA, Bernard A, Girard C. Comparison between systemic analgesia, continuous wound catheter analgesia and continuous thoracic paravertebral block: a randomised, controlled trial of postthoracotomy pain management. Eur J Anaesthesiol. 2012 Nov;29(11):524-30. doi: 10.1097/EJA.0b013e328357e5a1. PMID 22914044
- [Background] Fibla JJ, Molins L, Mier JM, Sierra A, Carranza D, Vidal G. The efficacy of paravertebral block using a catheter technique for postoperative analgesia in thoracoscopic surgery: a randomized trial. Eur J Cardiothorac Surg. 2011 Oct;40(4):907-11. doi: 10.1016/j.ejcts.2010.12.043. Epub 2011 Feb 11. PMID 21316259
- [Background] Helms O, Mariano J, Hentz JG, Santelmo N, Falcoz PE, Massard G, Steib A. Intra-operative paravertebral block for postoperative analgesia in thoracotomy patients: a randomized, double-blind, placebo-controlled study. Eur J Cardiothorac Surg. 2011 Oct;40(4):902-6. doi: 10.1016/j.ejcts.2011.01.067. Epub 2011 Mar 5. PMID 21377888
- [Background] Kaya FN, Turker G, Mogol EB, Bayraktar S. Thoracic paravertebral block for video-assisted thoracoscopic surgery: single injection versus multiple injections. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):90-4. doi: 10.1053/j.jvca.2011.09.008. Epub 2011 Nov 4. PMID 22055006
- [Background] Komatsu T, Sowa T, Takahashi K, Fujinaga T. Paravertebral block as a promising analgesic modality for managing post-thoracotomy pain. Ann Thorac Cardiovasc Surg. 2014;20(2):113-6. doi: 10.5761/atcs.oa.12.01999. Epub 2013 Feb 28. PMID 23445804
- [Background] Mackay, J. H., & Gray, S. J. (2013). Principles and Practice of Anesthesia for Thoracic Surgery. British Journal of Anaesthesia, 110(5), 857-858.
- [Background] Richardson J, Sabanathan S, Jones J, Shah RD, Cheema S, Mearns AJ. A prospective, randomized comparison of preoperative and continuous balanced epidural or paravertebral bupivacaine on post-thoracotomy pain, pulmonary function and stress responses. Br J Anaesth. 1999 Sep;83(3):387-92. doi: 10.1093/bja/83.3.387. PMID 10655907
- [Background] Shelley B, Macfie A. Where now for thoracic paravertebral blockade? Anaesthesia. 2012 Dec;67(12):1317-20. doi: 10.1111/j.1365-2044.2012.07310.x. No abstract available. PMID 23130723
- [Background] Slater, B., & Frost, E. A. (2012). Pain Management After Thoracic Surgery.Topics in Pain Management, 28(3), 1-8.
- [Background] Yoshida T, Fujiwara T, Furutani K, Ohashi N, Baba H. Effects of ropivacaine concentration on the spread of sensory block produced by continuous thoracic paravertebral block: a prospective, randomised, controlled, double-blind study. Anaesthesia. 2014 Mar;69(3):231-9. doi: 10.1111/anae.12531. Epub 2014 Jan 21. PMID 24447266
- [Background] Yoshioka M, Mori T, Kobayashi H, Iwatani K, Yoshimoto K, Terasaki H, Nomori H. The efficacy of epidural analgesia after video-assisted thoracoscopic surgery: a randomized control study. Ann Thorac Cardiovasc Surg. 2006 Oct;12(5):313-8. PMID 17095972
- [Result] Yeap YL, Wolfe JW, Backfish-White KM, Young JV, Stewart J, Ceppa DP, Moser EAS, Birdas TJ. Randomized Prospective Study Evaluating Single-Injection Paravertebral Block, Paravertebral Catheter, and Thoracic Epidural Catheter for Postoperative Regional Analgesia After Video-Assisted Thoracoscopic Surgery. J Cardiothorac Vasc Anesth. 2020 Jul;34(7):1870-1876. doi: 10.1053/j.jvca.2020.01.036. Epub 2020 Jan 25. PMID 32144059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group #1 | Group #2 | Group #3
Started | 53 | 47 | 47
Completed | 40 | 40 | 40
Not Completed | 13 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- US Guided Single Shot Paravertebral Block: group 1- US Guided Single Shot Paravertebral Block
  US Guided Single Shot Paravertebral Block (0.2% ropivicaine infusion): Single shot paravertebral block will be placed under ultrasound guidance at the thoracic region prior to surgery.
- US Guided Paravertebral Catheter: group 2- US Guided Paravertebral Catheter
  US Guided Paravertebral Catheter (0.2% ropivicaine bolus): Paravertebral catheter will be placed under ultrasound guidance at the thoracic region prior to surgery.
- Thoracic Epidural: group 3- Thoracic Epidural
  Thoracic Epidural (0.125% bupivicaine/hydromorphone): Epidural catheter will be placed in the thoracic region prior to surgery.
- Total: Total of all reporting groups
Arm/Group | US Guided Single Shot Paravertebral Block | US Guided Paravertebral Catheter | Thoracic Epidural | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.5 [48.5 to 70] | 62 [45.5 to 69.5] | 61 [52 to 70] | 62 [48 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 15 | 60
  Male | 16 | 19 | 25 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 40 | 40 | 40 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 4 | 1 | 13
  White | 32 | 33 | 39 | 104
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 40 | 120
height [Median (Inter-Quartile Range); unit: Centimeter] | 171 [162 to 177.8] | 167.6 [165 to 173.9] | 173.5 [161.3 to 179.3] | 170 [162 to 177.9]
weight [Median (Inter-Quartile Range); unit: Kilogram] | 88.4 [72.2 to 105] | 77.7 [67 to 90.4] | 87.3 [65.8 to 106.7] | 84.1 [67.1 to 102.1]

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study Will be VAS Pain Score at 24 Hours
Description: The VAS score will be taken with both rest and movement (knee flexion) and will be measured by a study team investigator using Visual Analog Scale (VAS). Using "units on a scale" of 1-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: Pain scores will be measured 24 hours after surgery.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | US Guided Single Shot Paravertebral Block | US Guided Paravertebral Catheter | Thoracic Epidural
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 4.0 [3.0 to 5.5] | 4.5 [2.5 to 6.0] | 3.0 [1.0 to 5.0]

2. Primary Outcome: The Primary Endpoint of This Study Will be VAS Pain Score at 48 Hours
Description: The VAS scores will be taken with both rest and movement (knee flexion) and will be measured by a study team investigator using Visual Analog Scale (VAS). Using"units on a scale" scale of 1-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: Pain scores will be measured 48 hours after surgery.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | US Guided Single Shot Paravertebral Block | US Guided Paravertebral Catheter | Thoracic Epidural
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 3.0 [1.0 to 5.0] | 4.0 [2.0 to 6.0] | 2.0 [1.0 to 4.0]

3. Secondary Outcome: Secondary Endpoint Includes Total Intravenous Opioid Consumption at 72 Hours
Description: Opioid consumption will be collected by a study team member post operatively up to 3 days per protocol time requirements
Time Frame: Opioid consumption will be measured at 1 hour post op, 24,48, and 72 hours post op. The total amount will be recorded.
Measure: Median (Inter-Quartile Range); unit: miligram morphine equivalent
Arm/Group | Group #1 | Group #2 | Group #3
Number analyzed (Participants) | 40 | 40 | 40
miligram morphine equivalent | 57 [18 to 96] | 35 [15 to 89] | 21.3 [7.5 to 45]

4. Other Pre Specified Outcome: Average Nausea Scores Over 72 Hours
Description: Nausea scores will be collected by a study team member post operatively up to 3 days per protocol. Nausea will be recorded as 0=none, 1=mild, 2=moderate, or 3=severe
Time Frame: Nausea scores will be documented at 1 hour post op, 24,48,and 72 hours after the surgery.The scores will then be averaged.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Group #1 | Group #2 | Group #3
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 0.27 [0 to 3] | 0.27 [0 to 3] | 0.29 [0 to 3]

5. Other Pre Specified Outcome: Average Sedation Scores Over 72 Hours
Description: Sedation scores will be documented by a study team member post operatively up to 3 days per protocol requirements. Determining if patient is 0=awake and alert, 1=quietly awake, 2=asleep and arousable, or 3=deep sleep.
Time Frame: Sedation scores will be documented at 1 hour post op, 24,48,and 72 hours after the sugery. The scores will then be averaged.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Group #1 | Group #2 | Group #3
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 0.38 [0 to 3] | 0.32 [0 to 3] | 0.22 [0 to 3]

6. Other Pre Specified Outcome: Subjects Overall Satisfaction Scores
Description: Subjects will be followed up at 24 hours post operatively by a study team member to document patient overall satisfaction scores. Score was recorded as 0=dissatisfied, 1=satisfied, 2=very satisfied.
Time Frame: post operatively at hour 24
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Group #1 | Group #2 | Group #3
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 0.89 [0 to 2] | 0.95 [0 to 2] | 1.33 [0 to 2]

7. Other Pre Specified Outcome: Subjects Overall Satisfaction Scores
Description: Subjects will be followed up at 48 hours post operatively by a study team member to document patient overall satisfaction scores. Scores will be recorded as 0=dissatisfied, 1=satisfied, 2=very satisfied.
Time Frame: post operatively at hour 48
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Group #1 | Group #2 | Group #3
Number analyzed (Participants) | 40 | 40 | 40
units on a scale | 1.19 [0 to 2] | 1.05 [0 to 2] | 1.32 [0 to 2]

ADVERSE EVENTS:
Time Frame: Participants were followed for 6 months after surgery. Any adverse event from surgery day till 6 months after surgery are documented.
Arm/Group | US Guided Single Shot Paravertebral Block | US Guided Paravertebral Catheter | Thoracic Epidural
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT03151434/Prot_SAP_001.pdf